CLINICAL TRIAL: NCT06399484
Title: Immediate Effect of Median Nerve Mobilization on Neural Conduction in Patients With Carpal Tunnel Syndrome: Randomized Clinical Trial
Brief Title: In Patients With Carpal Tunnel Syndrome, Median Nerve Conduction is Evaluated After Nerve Mobilizations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena Bueno Gracia, Physiotherapist, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23/437
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization group (Experimental): Manual mobilizations of the median nerve.
  Interventions: Other: Manual mobilizations of the median nerve
- Placebo group (Placebo Comparator): wrist movements no producing sliding of the median nerve
  Interventions: Other: Wrist movements

INTERVENTIONS:
Other: Manual mobilizations of the median nerve — Slippage of the median nerve in the wrist: the subject's starting position (P0) will be recumbent supine with the cervical spine in a neutral position, the shoulder girdle in neutral position, 30º of glenohumeral abduction in neutral rotation, 90º of elbow flexion, prone-supination of the neutral forearm, wrist and fingers in neutral position. From this position the movements will be 1) Glenohumeral abduction up to 90º; 2) Glenohumeral external rotation to the frontal plane; 3) Supination of the forearm; 4) Extension of the wrist and fingers; 5) Elbow extension. This position is will combine with an ipsilateral cervical inclination (distal sliding). The proximal slide is carried out bringing the fingers of the hand towards the flexion while performing a contralateral cervical tilt.
  Median nerve tension: the starting position and movements are the same described above but this time it will be done with contralateral cervical tilt.
  Arms: Neural mobilization group
Other: Wrist movements — Movements of the wrist joint will be performed as a placebo treatment
  Arms: Placebo group

SUMMARY:
This project is linked to the line of research on carpal tunnel syndrome, of the PhysiUZerapy research group, belonging to the University of Zaragoza. Within this line, the biomechanical and physiological effect of the proposed technique has been investigated, both in healthy subjects, in cadavers and in patients with carpal tunnel syndrome (CTS), resulting in the reading of 2 doctoral theses, the publication of 9 articles in high-impact journals. and the patent for a splint for the treatment of pathology. This project aims to provide information that is still lacking on the immediate effect of these techniques in patients with CTS. For this, there will be three groups of patients from the Lozano Blesa University Clinical Hospital distributed randomly. In two of the groups, sliding and neural tension techniques will be carried out (case group). The remaining group (control group) will be taken as a reference by performing a placebo treatment. Before and after carrying out these techniques, electrophysiological data will be collected to be able to compare them. This comparison is based on highlighting the differences between the data before the techniques and after, as well as between the case group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years
* Present carpal tunnel syndrome diagnosed by electroneurogram
* Have understanding and communication skills
* Give consent to participate in the study

Exclusion Criteria:

* Have received previous surgery on the hand or wrist
* Present a severe limitation of movement in any of the joints of the affected upper limb
* Not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Distal motor latency (APB) (ms) | Before and immediately after the intervention
Motor amplitude (APB) (mV) | Before and immediately after the intervention
Median motor velocity (m/s) | Before and immediately after the intervention
Median sensory conduction (digit II) (13 cm) (m/sec) | Before and immediately after the intervention
Sensory amplitude (µV) | Before and immediately after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT06399484/ICF_000.pdf